CLINICAL TRIAL: NCT03740880
Title: Pilot Study: Optimal Trigger Time in Advanced Maternal Age Patients With Low AMH
Brief Title: Trigger Time in Advanced Maternal Age Patients With Low AMH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient data
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1810-ABU-067-HF
Record Dates: First submitted 2018-11-12; First posted 2018-11-14 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: the Number of Mature Oocytes
Keywords: ICSI; early trigger; poor ovarian responders; low AMH

STUDY DESIGN:
Intervention Model Description: Two groups: 1 groups of patients receiving an early trigger (14mm), the other group receiving a late trigger (17mm)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Late trigger (Active Comparator): dual trigger (10.000 IU hCG i.m. and 0.3 mg Deca) once the leading follicle is 17 mm
  Interventions: Other: Dual trigger
- Early trigger (Experimental): dual trigger (10.000 IU hCG i.m. and 0.3 mg Deca) once the leading follicle is 14 mm
  Interventions: Other: Dual trigger

INTERVENTIONS:
Other: Dual trigger — dual trigger: 10.000 IU hCG i.m. and 0.3 mg Deca

SUMMARY:
The investigators want to verify if advanced maternal age patients with a low Anti-Müllerian hormone (AMH) level may benefit from an early trigger time (compared to a late trigger).

DETAILED DESCRIPTION:
During assisted reproduction, patients are stimulated in order to achieve a multifollicular development. The final step in this stimulation process is "the trigger" that will induce the final maturation of the oocytes. This timing is historically put once at least one follicle of 16-17 mm is obtained.

When looking at poor ovarian responder (POR) patients (characterized by a low AMH), the investigators observe shorter menstrual cycles and thus it is thought that the oocyte selected for ovulation, will also mature faster. This observation may indicate that POR patients potentially do not benefit from a trigger performed once a leading follicle of 17 mm is present, but rather from an earlier trigger.

The main objective is to analyse if an early trigger (leading follicle of 14 mm) results in the same maturation rate in POR patient as compared to a late trigger (17 mm). As the embryos will be cultured in a time lapse imaging system, annotations on the developmental kinetics can be made and the differences in fertilization rate and embryo development can be analysed as secondary outcome parameter. On top of this, patients will undergo a genetic testing of their embryos and this genetic analysis , together with the mtDNA copy number will also be compared between patients with early or late trigger. Euploid blastocysts will be transferred in subsequent frozen embryo transfer (FET) cycles and give an indication on the clinical outcome between IVF and ICSI.

ELIGIBILITY:
Inclusion Criteria:

* • POR defined according to the Bologna criteria:

  * AMA: ≥40 years and AMH <1.1 ng/ml
  * Previous poor ovarian response with maximum 3 cumulus oocyte complexes retrieved after conventional stimulation
  * Antral follicle count < 5-7

    * Cycling patients
    * Fresh ejaculates
    * ICSI
    * BMI 19-32 kg/m2
    * Ovarian stimulation protocol: Antagonist HMG 450 IU to ensure all receptors are covered and to ensure maximum recruitment. Dose adjustments can be made after 5 days of stimulation
    * Type of trigger for final oocyte maturation: dual trigger: 10.000 IU hCG i.m. and 0.3 mg Deca
    * Couples requesting preimplantation genetic testing (for aneuploidies) of their embryos
    * Follicular measurements should be performed at IVI RMA Fertility, Abu Dhabi, UAE: a single operator will perform the ultrasound for the final measurement before trigger. Recruitment can be done by all physicians
    * Only patients with an oral contraceptive pill (OCP) pretreatment to synchronize follicular development:
  * 2 weeks OCP followed by
  * a wash out of 5 days (without OCP) followed by

    * o start stimulation
    * Basal hormone profile (FSH, LH, E2, P4) measured between day 1-3 at IVIRMA Fertility, Abu Dhabi, UAE
  * FSH <15 IU
  * E2 <50 pg/ml
  * P <1ng/ml

    * Only the Arab population
    * Oocyte retrieval: 36 hours after trigger
    * PGT-A

Exclusion Criteria:

* If follicular measurement before randomization shows a leading follicle ≥ 13mm
* IVF
* History of:

  * Endometriosis AFS>2
  * Chemotherapy/radiotherapy
  * Ovarian surgery (iatrogenic)
  * Cyst puncture in the last three months
* Sonographic finding of:

  * Hydrosalpinx
  * Ovarian cyst
* Testicular samples and frozen ejaculates
* If patients are pre-screened at the start of stimulation but no follicular development is observed, patients will not be randomized
* Asynchronized follicular development at the moment of randomization: if the leading follicle is >3 mm lager than the smaller follicles.
* All other hormonal pretreatments (except OCP) and all patients without hormonal pretreatment

Ages: 40 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only female patients can undergo an ovarian stimulation protocol
Enrollment: 1 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
the number of mature oocytes | 1 day
  A mature oocyte is defined as an oocyte that has extruded his first polar body and this mature oocyte is ready to be fertilized by the participants sperm.

SECONDARY OUTCOMES:
Maturation rate | 1 day
  The maturation rate is defined as the number of mature oocytes obtained per cumulus complex retrieved for the participants.A mature oocyte is defined as an oocyte that has extruded his first polar body and this mature oocyte is ready to be fertilized by the participants sperm.
Fertilization rate | 1 day
  Fertilization is calculated on all mature oocytes or on all complexes obtained after oocyte retrieval. The fertilization rate is assessed by the presence of a male and a female pronucleus 16-20 hours post fertilization. If the oocyte is fertilized, the outcome is positive, if the oocyte is not fertilized, the outcome is negative.
Embryo development up to day 3 | 3 days
  For all normally fertilized oocytes the further development will be assessed as the embryos are cultured in a time lapse system. This system takes pictures of the embryos every 20 minutes which shows the development of the embryo like a movie: every time that a cell divides, the hour at which it divides will be registered in the time lapse system. For each cell division, specific time frames have been described that link the embryo to develop into a blastocyst or that increases the chance of implantation. The embryo will be evaluated on day 3 and will receive an embryo score that is based on the number of cells, the appearance of the cells, fragmentation and embryo dysmorphisms. These will divide the embryo quality into 4 categories with category 1 being the highest quality and category 4 being the lowest quality. The more fragmentation and the higher the degree of dysmorphisms, the more the quality will shift to category 4
Blastulation rate | 7 days
  A blastocyst is an embryo in which a cavity is visible on day 5 of the embryo development. If the cavity is present the outcome is positive, if the cavity is absent, the outcome is negative The complete process in which the development of one embryo is followed from the day of injection up until day 7 is called the preimplantation development
Embryo development up to day 5 | 7 days
  On day 5 of development, a score is given to every embryo. This is based on the presence or absence of a cavity, the number of cells and how tight the cells are packed. The more cells, the higher the grade, if less cells are present, the grade is lower. Based on these parameters, a final grade is calculated (3 grades) with grade 1 being the highest score.
Morphokinetic development | 7 days
  As embryos are cultured in a time lapse imaging system, pictures will be taken every 20 minutes to follow the development. Each time that the embryos divides, the timing will be registered in the database. Like this, every division made by every embryo is recorded: the time the embryo needs to go from 1 cell to 2 cells, from 2 cells to 3 cells and so on.
Ploidy state: euploid or aneuploid | 7 days
  Trophectoderm biopsy performed between day 5-7 of preimplantation development. These cells will be genetically tested to see if the correct number of chromosomes are present. Euploid embryos can be used for the patient, aneuploid embryos cannot be used for the patient.
Mitoscore value: ranges from 10-1500 | 7 days
  The trophectoderm biopsy sample is used to calculate a value indicating the mitochondrial DNA present in the biopt. Lower values are known to be linked to higher implantation rates of the corresponding blastocyst. Higher values have been correlated to aneuploidy.
Pregnancy outcome | 3 months
  Pregnancy outcomes from the frozen embryo transfers: blood samples will be taken and the level of beta-hCG will be measured to define a pregnancy or no pregnancy. A pregnancy is defined as the best oucome. In case a pregnancy is obtained, the patient will come for an ultrasound scan between week 7-12 to checke the presence of a gestational sac and the presence of a fetal heart beat. The presence of a fetal heart beat is defined as a positive outcome, the absence is defined as a negative outcome.

OTHER OUTCOMES:
Controlled ovarian stimulation: dosage | 2 weeks
  In order to stimulate multiple follicular development, patients will be stimulated with fixed doses of hormones. The total dosage of hormones used will be registered.
Controlled ovarian stimulation: days of stimulation | 2 weeks
  In order to stimulate multiple follicular development, patients will be stimulated with fixed doses of hormones. Once the follicular development is optimal (based on the number of follicles and the corresponding hormonal values) the patient can be triggered for final oocyte maturation. The total number of days needed during this stimulation will be registered.
Controlled ovarian stimulation: hormonal profile | 2 weeks
  During the stimulation, the hormonal profile of every patient will be measured (estrogens, luteinizing hormone, progesterone): these blood values will be compared to the number of follicles that are measured in the participants and the combination of the three blood values should correspond to the sizes and numbers of follicles measured in the participants.
Controlled ovarian stimulation: measurement of follicles | 2 weeks
  During the stimulation, the follicles present in the participants will grow steadily and the size of the follicles will be measured on a regular basis to ensure a good development (in combination with the hormonal profile). These follicles will be measured by vaginal echography.
Mean menstrual cycle length | 3 months
  the last three months before the stimulation start, the participant will be asked the length of her last three menstrual cycles. The average of the three will give the value needed.

CONTACTS AND LOCATIONS:
Overall Officials: Neelke De Munck, PhD, Principal Investigator — IVIRMA Abu Dhabi
Locations (1):
- IVI RMA Abu Dhabi, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided
Information regarding primary and secondary outcome measures will only be shared with researchers from the clinic, involved in the study.

REFERENCES:
- [Result] Haahr T, Esteves SC, Humaidan P. Individualized controlled ovarian stimulation in expected poor-responders: an update. Reprod Biol Endocrinol. 2018 Mar 9;16(1):20. doi: 10.1186/s12958-018-0342-1. PMID 29523204
- [Result] Oudendijk JF, Yarde F, Eijkemans MJ, Broekmans FJ, Broer SL. The poor responder in IVF: is the prognosis always poor?: a systematic review. Hum Reprod Update. 2012 Jan-Feb;18(1):1-11. doi: 10.1093/humupd/dmr037. Epub 2011 Oct 10. PMID 21987525
- [Result] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Result] Beckers NG, Macklon NS, Eijkemans MJ, Fauser BC. Women with regular menstrual cycles and a poor response to ovarian hyperstimulation for in vitro fertilization exhibit follicular phase characteristics suggestive of ovarian aging. Fertil Steril. 2002 Aug;78(2):291-7. doi: 10.1016/s0015-0282(02)03227-2. PMID 12137865